CLINICAL TRIAL: NCT04423198
Title: HEAD Injury Serum Markers and Multi-modalities for Assessing Response to Trauma II
Brief Title: HEAD Injury Serum Markers and Multi-modalities for Assessing Response to Trauma
Acronym: HeadSMART II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BRAINBox Solutions Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN01001
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: TBI, mTBI
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — Mental Status and Dementia Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen Samples for the analysis of biomarkers include:
  1. Serum
  2. RNA
  3. Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Target Condition: Subjects presenting to the Emergency Department (ED) or Urgent Care (UC) with a blunt head trauma
  Interventions: Behavioral: Cognitive Assessment; Behavioral: Patient Reported Neurological Outcome Assessments; Procedure: Blood Draw
- Trauma Control: Subjects presenting to the ED or UC requiring an Xray but do not have a head trauma
  Interventions: Behavioral: Cognitive Assessment; Behavioral: Patient Reported Neurological Outcome Assessments; Procedure: Blood Draw
- Healthy Control: Subjects that are healthy and not taking any prescription medications
  Interventions: Behavioral: Cognitive Assessment; Procedure: Blood Draw

INTERVENTIONS:
Behavioral: Cognitive Assessment — Self administered cognitive battery
Behavioral: Patient Reported Neurological Outcome Assessments — Standard neurocognitive and neuropsychological tests
  Groups: Target Condition; Trauma Control
Procedure: Blood Draw — Specimen collection of whole blood, serum, RNA

SUMMARY:
The goal of HeadSMART II (HEAD injury Serum markers and Multi-modalities for Assessing Response to Trauma II) is to develop an In-Vitro Diagnostic, the BRAINBox TBI test, to aid in the diagnosis and prognosis of patients with mild traumatic brain injury, by incorporating blood biomarkers, clinical assessments, and tools to measure associated neurocognitive impairments.

DETAILED DESCRIPTION:
This study proposes to collect data using a multi-modality approach including blood biomarkers, clinical assessments, neurocognitive performance, and neuropsychological characteristics, to identify subjects with a mild Traumatic Brain Injury (TBI) and their likelihood of chronic symptoms.

This is an observational study with an expectation of enrolling up to 2000 subjects. These subjects will include the intended use population, subjects presenting to the Emergency Department or Urgent Care with a blunt head trauma. Data will be collected across four time points, T=0, 14 days, 30 days and 90 days, to allow for building and validating the algorithms for both diagnosis and prognosis claims.

Control populations, healthy and trauma only (no head trauma) will be included for assay development. Data will be collected for these groups at T=0 and 14 days (trauma control only).

ELIGIBILITY:
Target Condition Subjects

Inclusion Criteria:

1. Age >=18 years
2. Ability to provide a blood sample; within 96 hours of injury
3. Ability to provide informed consent. Consent may be obtained with assistance of a legally authorized representative (LAR)
4. Must present to the Emergency Department (ED) or Urgent Care (UC) with a blunt head trauma

Exclusion Criteria:

1. Glasgow Coma Scale (GCS) score < 13, as presented in ED at time of screening
2. Need for general anesthesia at the time of presentation in the ED
3. Diagnosed dementia requiring assistance for daily living
4. Any head trauma requiring medical attention from a physician within the last 6 months
5. Received chemotherapy or radiation within the last year
6. History of stroke with disabling outcomes, brain tumor, epilepsy or intracranial surgery/hemorrhage
7. Psychiatric hospitalization in the last 90 days
8. Blood transfusion within the prior 4 weeks
9. Non-working telephone number
10. Current participant in an interventional clinical trial
11. Cannot perform study tasks on an iPad (e.g. not wearing corrective lenses necessary to read, inability to use both hands)
12. Subject considered unsuitable for participation in this clinical trial by PI, treating clinician or research study staff

Control Subjects

Inclusion:

1. Age >=18 years
2. Ability to provide a blood sample; (For Trauma Controls (TC's) within 96 hours of injury)
3. Ability to provide informed consent. (For TC's consent may be obtained with assistance of a legally authorized representative (LAR)
4. Presents to the Emergency Department or Urgent Care with at least one injury requiring an X-Ray (TC's only)
5. Healthy and not taking prescription medications (Healthy Controls (HC's) only)

Exclusion:

1. Head trauma or symptoms with head trauma at presentation
2. Head trauma requiring medical attention from a physician within the last 6 months
3. Internal organ injury (e.g. liver laceration, pulmonary contusion, spinal cord injury) that requires inpatient hospitalization
4. Need for general anesthesia at the time of presentation in the ED
5. Diagnosed dementia requiring assistance for daily living
6. Received chemotherapy or radiation within the last year
7. History of stroke with disabling outcomes, brain tumor, epilepsy or intracranial surgery/hemorrhage
8. Psychiatric hospitalization in the last 90 days
9. Blood transfusion within the prior 4 weeks
10. Non-working telephone number
11. Current participant in an interventional clinical trial
12. Cannot perform study tasks on an iPad (e.g. not wearing corrective lenses necessary to read, inability to use both hands)
13. Subject considered unsuitable for participation in this clinical trial by PI, treating clinician or research study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to the Emergency Department or Urgent Care with a blunt head trauma.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of mild traumatic brain injury diagnosis using the BRAINBox TBI Test compared to the Expert Clinical Diagnosis | 30 days
  Sensitivity and specificity of the diagnosis as compared to a clinical diagnosis by an expert committee
Determine the risk stratification of having symptoms at 14, 30 and 90 days, for subjects with mild traumatic brain injury using the BRAINBox TBI Test results. | up to 90 days
  Sensitivity and specificity of the risk for chronic symptoms as compared to the post-concussion symptoms at predefined time points

CONTACTS AND LOCATIONS:
Overall Officials: Frank Peacock, MD, Principal Investigator — Baylor College of Medicine
Locations (11):
- United States (11):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Detroit Receiving, Detroit, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook Medicine, Stony Brook, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - John Peter Smith (JPS) Health Network, Fort Worth, Texas
  - Baylor College of Medicine/Ben Taub, Houston, Texas
  - Baylor College of Medicine/St. Luke's Medical Center, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Undecided